CLINICAL TRIAL: NCT06096012
Title: Don't Treat Ghosts: Anti-MRSA Antibiotics in Osteomyelitis Without Identified MRSA
Brief Title: Don't Treat Ghosts Anti-MRSA Antibiotics in Osteomyelitis Without Identified MRSA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 025.PHA.2023.A
Record Dates: First submitted 2023-10-17; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-08

CONDITIONS: Osteomyelitis
MeSH Terms: conditions — Osteomyelitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Anti-MRSA therapy — chart review to determine the clinical outcomes of patients with osteomyelitis who were placed on definitive anti-MRSA treatment, despite no identified MRSA cultures.
  Other Names: Anti-MRSA Antibiotics

SUMMARY:
Osteomyelitis is described as infection and inflammation of the long bone or bone marrow, often due to an open wound, operation, or invasive trauma.1 It is invasive and involves hematogenous seeding or contiguous spread of the infectious organism

DETAILED DESCRIPTION:
This disease can be classified by location of infection, extent of spread, chronicity, and source of infection.3,4 Osteomyelitis can be caused by a variety of organisms, most commonly gram-positive staphylococci.

Osteomyelitis is associated with a high rate of relapse, high disease burden, and high health care costs.3 Following confirmation of disease via imaging and histopathologic examination, treatment consists of antibiotic therapy and, often, surgical intervention.3,5,6 Treatment with antibiotic therapy is often administered for 4-6 weeks when surgical intervention is not performed.6 Antibiotic selection should be guided by microbiology and antimicrobial susceptibilities.4 Thirty to sixty percent of osteomyelitis cases are caused by Staphylococcus aureus.

ELIGIBILITY:
Inclusion Criteria:

* • Admission to any MHS hospital between April 1, 2017 and April 1, 2023

  * > 18 years of age
  * Documented osteomyelitis location of the lower limb via ICD-10 code
  * Documented imaging of lower limb osteomyelitis during index admission
  * Planned intravenous (IV) antibiotics for at least 4 weeks

Exclusion Criteria:

* • IV antibiotics for less than 24 hours inpatient

  * Planned surgical intervention documented at admission
  * Patients receiving monotherapy with an anti-MRSA agent
  * Positive MRSA culture during index admission
  * Current outpatient antibiotic use on index admission
  * Repeated hospital admission during study period

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to any MHS hospital between April 1, 2017 and April 1, 2023
  * > 18 years of age
  * Documented osteomyelitis location of the lower limb via ICD-10 code
  * Documented imaging of lower limb osteomyelitis during index admission
  * Planned intravenous (IV) antibiotics for at least 4 weeks
Sampling Method: Non-Probability Sample
Enrollment: 365 (Estimated)
Dates: Start 2023-06-23 (Actual); Primary Completion 2024-06-23 (Estimated); Study Completion 2024-06-23 (Estimated)

PRIMARY OUTCOMES:
Comparison of treatment | 180 Days
  the comparison of treatment failure between anti-MRSA therapy and no anti-MRSA therapy defined as a composite of hospital readmission for osteomyelitis within 180 days of antibiotic initiation

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Crotty, PharmD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
The PI is committed to disseminate research results in a timely fashion. Sharing of data generated by this project will be carried out through presentation at scientific meetings and/or publication in Open Access Journals.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 2 years
Access Criteria: Clinical trials portal or CRI MHS

REFERENCES:
- [Background] Jha Y, Chaudhary K. Diagnosis and Treatment Modalities for Osteomyelitis. Cureus. 2022 Oct 26;14(10):e30713. doi: 10.7759/cureus.30713. eCollection 2022 Oct. PMID 36439590
- [Background] Hirschfeld CB, Kapadia SN, Bryan J, Jannat-Khah DP, May B, Vielemeyer O, Esquivel EL. Impact of diagnostic bone biopsies on the management of non-vertebral osteomyelitis: A retrospective cohort study. Medicine (Baltimore). 2019 Aug;98(34):e16954. doi: 10.1097/MD.0000000000016954. PMID 31441894